CLINICAL TRIAL: NCT05982938
Title: Early Access Program (EAP) for Danicopan as Add-on Treatment to SOLIRIS® or ULTOMIRIS® in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Who Have Clinically Significant Extravascular Hemolysis (csEVH)
Brief Title: Danicopan Early Access Program
Status: Available | Type: Expanded Access
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D7332R00001
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria; PNH; Extravascular Hemolysis
Keywords: paroxysmal nocturnal hemoglobinuria; PNH; component 5 inhibitors; C5i; intravascular hemolysis; IVH; anemia; EVH; extravascular hemolysis
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemolysis; Anemia | interventions — danicopan

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Danicopan — Participants will receive 150 mg danicopan three times per day (TID) orally as an add-on to a background C5i therapy (SOLIRIS® or ULTOMIRIS®). Participants may be dose-escalated to 200 mg TID based on safety and clinical effect.
  Other Names: ALXN2040

SUMMARY:
This is an EAP, designed to provide early access to danicopan for participants with PNH experiencing clinically significant EVH who have failed, not tolerated, or are unable to receive other approved treatments; in the Treating Physician's opinion, the participant is not eligible for or is not able to participate in an ongoing clinical trial of danicopan or a comparable treatment; and according to the Treating Physician, the benefit of danicopan treatment outweighs the potential risks.

ELIGIBILITY:
Key Inclusion Criteria

* Male or female, aged 18 years and older
* Diagnosed with PNH with clinically significant EVH as defined by anemia (Hgb ≤ 9.5 g/dL) with absolute reticulocyte count ≥ 120 × 109/L.
* Currently receiving treatment with SOLIRIS® or ULTOMIRIS® for at least 6 months prior to initiation of danicopan treatment.
* Platelet count ≥ 30,000/µL without the need for platelet transfusions.
* Absolute neutrophil counts ≥ 500/µL.
* Vaccinated against N meningitidis.

Key Exclusion Criteria

* Participants who are nursing or pregnant (or women who are planning to become pregnant during treatment with danicopan).
* Laboratory abnormalities at screening, as follows:
* Alanine aminotransferase (ALT) > 2 × upper limit of normal (ULN)
* Direct bilirubin > 2 × ULN, with the exception of:

  * participants with increased bilirubin due to EVH in the opinion of the Treating Physician or
  * participants with documented Gilbert's syndrome
* Active bacterial or viral infection, a body temperature > 38°C on 2 consecutive daily measures, evidence of other infection, or history of any febrile illness within 14 days prior to initiating danicopan treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult